CLINICAL TRIAL: NCT00006035
Title: An Open Label Lesion Controlled Study of Electroporation Therapy (EPT) for the Treatment of Cutaneous Metastatic Melanoma Using the Genetronics, Inc. Medpulser System and Bleomycin
Brief Title: Bleomycin With or Without Electroporation Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068050; MCC-11883; GENETR-EPT-9706001; MCC-IRB-5219; NCI-G00-1811
Record Dates: First submitted 2000-07-05; First posted 2004-06-21 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2000-11

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Bleomycin; Electroporation Therapies

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: electroporation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Electroporation therapy may enhance the ability of chemotherapy drugs to enter tumor cells. Combining chemotherapy with electroporation therapy may kill more tumor cells.

PURPOSE: Randomized phase I trial to compare the effectiveness of bleomycin with or without electroporation therapy in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the objective tumor response rate of patients with stage III or IV melanoma when treated with intratumoral bleomycin with or without electroporation therapy. II. Determine the safety of electroporation therapy in these patients. III. Compare the time to heal with these treatments in these patients. IV. Compare the duration of lesion response with these treatments in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive bleomycin intratumorally on day 1. Arm II: Patients receive bleomycin intratumorally followed by electroporation therapy intratumorally on day 1. Treatment continues every 4 weeks in the absence of unacceptable toxicity. Patients in arm I with progressive disease after 1 course of treatment may be crossed over to arm II. Patients are followed at 4 and 6 months after final treatment.

PROJECTED ACCRUAL: A total of 20 patients (10 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV melanoma Progressive disease defined by: Stage III Inoperable due to number of lesions (greater than 5 nodules) OR Recurrence after surgical excision Stage IV Failed to respond to immunotherapy or chemotherapy OR Immunotherapy or chemotherapy contraindicated Bidimensionally measurable disease At least 2 lesions accessible to electroporation electrode

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Greater than 6 months Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine clearance at least 35 mL/min Cardiovascular: No cardiac pacemakers or implantable defibrillators No history of severe cardiac arrhythmia No myocardial infarction in past 6 months Pulmonary: No significant pulmonary fibrosis or other severe pulmonary pathology Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No clinical or bacteriological evidence of active infection No known hypersensitivity to bleomycin including shock, uncontrolled hypothermia, prurit or prurit type toxidermia, Raynaud's syndrome, or digital gangrene No known sensitivity to lidocaine

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Concurrent systemic immunotherapy allowed if disease is stable or progressing at time of study entry after at least 8 weeks of treatment Chemotherapy: See Disease Characteristics At least 12 weeks since prior intralesional chemotherapy Concurrent systemic chemotherapy allowed if disease is stable or progressing at time of study entry after at least 8 weeks of treatment Must not have previously exceeded or will exceed on this study a cumulative dose greater than 400 U of bleomycin Endocrine therapy: Not specified Radiotherapy: At least 12 weeks since prior local radiotherapy to study lesion Surgery: See Disease Characteristics At least 12 weeks since prior local surgery to study lesion Other: At least 12 weeks since prior local cryotherapy to study lesion At least 4 weeks since prior investigational drugs or devices No other concurrent investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C. DeConti, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States